CLINICAL TRIAL: NCT01535729
Title: Erlotinib (Tarceva®) in Routine Clinical Practice in Patients With Advanced Non Small Cell Lung Cancer (NSCLC) After Failure of at Least One Prior Chemotherapy Regimen With Focus on the Elderly Patient.
Brief Title: An Observational Study of Tarceva (Erlotinib) in Elderly Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML23023
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate the efficacy and safety of Tarceva (erlotinib) in elderly patients with advanced non-small cell lung cancer (NSCLC) after failure of at least one prior chemotherapy regimen. Data of patients treated with Tarceva in routine clinical practice will be collected for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, > 65 years of age
* Locally advanced or metastatic non-small cell lung cancer (Stage IIIb or IV)
* Failure of at least one prior standard platinum-based chemotherapy

Exclusion Criteria:

* Age < 65 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with advanced non-small cell lung cancer after first-line platinum-based chemotherapy
Sampling Method: Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Nuremberg, Germany

REFERENCES:
- [Derived] Brueckl WM, Achenbach HJ, Ficker JH, Schuette W. Erlotinib treatment after platinum-based therapy in elderly patients with non-small-cell lung cancer in routine clinical practice - results from the ElderTac study. BMC Cancer. 2018 Mar 27;18(1):333. doi: 10.1186/s12885-018-4208-x. PMID 29587656

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-small Cell Lung Cancer (NSCLC) Elderly Participants: Elderly Participants (greater than or equal to [≥] 65 years) with locally advanced or metastatic NSCLC, on erlotinib (Tarceva®) prescribed in accordance with the terms of the marketing authorization, were observed for maximum of 12 months.
Period: Overall Study
Arm/Group | Non-small Cell Lung Cancer (NSCLC) Elderly Participants
Started | 465
Treated | 385
Completed | 49
Not Completed | 416
Not completed — Withdrawal by Subject | 2
Not completed — Disease progression | 230
Not completed — Discontinued treatment | 25
Not completed — Lost to Follow-up | 8
Not completed — Death | 52
Not completed — Other | 19
Not completed — Did not sign informed consent | 1
Not completed — No previous chemotherapy | 33
Not completed — NSCLC grade IV histology not confirmed | 20
Not completed — Protocol Violation | 11
Not completed — Screening failure | 1
Not completed — Not treated | 9
Not completed — No participant record available | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF), included participants who received at least one dose of Tarceva®.
Groups:
- NSCLC Elderly Participants: Elderly Participants (≥ 65 years) with locally advanced or metastatic NSCLC, on erlotinib (Tarceva®) prescribed in accordance with the terms of the marketing authorization, were observed for maximum of 12 months.
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.66 (5.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 258

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Alive 1 Year After Start of Treatment
Description: Overall survival was defined as the time from the date of first medication to the date of death from any cause. If death was not observed during the study, survival time was censored at the last day of observation (latest at the end of study after one year). Overall percentage of participants who were alive 1 year after study treatment and those based on the factor of age (65-69, 70-74, 75-79, ≥ 80 years) were reported.
Time Frame: Year 1
Population: SAF
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Overall | 30.6 [25.2 to 36.0]
  65-69 years | 26.6 [16.8 to 36.3]
  70-74 years | 29.8 [20.6 to 39.0]
  75-79 years | 37.2 [26.3 to 48.2]
  ≥ 80 years | 25.6 [9.0 to 42.3]

2. Secondary Outcome: Median Overall Survival: Age
Description: Overall Survival was defined as the time from the date of first medication to the date of death from any cause. If death was not observed during the study, survival time was censored at the last day of observation (latest at the end of study after one year). Overall Survival was analyzed by means of Kaplan-Meier Methods. Median survival based on the factor of age (65-69, 70-74, 75-79, ≥80 years) were reported.
Time Frame: From Baseline then every 3 months from Month 3 until death (Maximum follow-up to Month 40)
Population: SAF
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
months
  65-69 years | 7.039 [5.033 to 8.717]
  70-74 years | 6.612 [5.164 to 8.125]
  75-79 years | 7.928 [6.118 to 11.349]
  ≥ 80 years | 6.020 [4.507 to 10.954]
Statistical Analysis 1: Comparison: NSCLC Elderly Participants; Comparison between 70-74 years and 65-69 years was reported. Parameter estimates, standard errors, Wald Chi-Squares, p-values, hazard ratios and confidence limits were based on a univariate Cox regression with factor age; Test type: Superiority or Other; p = 0.756, Wald Chi-Squares; Hazard Ratio (HR) = 0.949, 95% CI 2-sided [0.684 to 1.318], Standard Error of Mean 0.167
Statistical Analysis 2: Comparison: NSCLC Elderly Participants; Comparison between 75-79 years and 65-69 years was reported. Parameter estimates, standard errors, Wald Chi-Squares, p-values, hazard ratios and confidence limits were based on a univariate Cox regression with factor age; Test type: Superiority or Other; p = 0.110, Wald Chi-Squares; Hazard Ratio (HR) = 0.744, 95% CI 2-sided [0.518 to 1.070], Standard Error of Mean 0.185
Statistical Analysis 3: Comparison: NSCLC Elderly Participants; Comparison between ≥ 80 years and 65-69 years was reported. Parameter estimates, standard errors, Wald Chi-Squares, p-values, hazard ratios and confidence limits were based on a univariate Cox regression with factor age; Test type: Superiority or Other; p = 0.829, Wald Chi-Squares; Hazard Ratio (HR) = 1.054, 95% CI 2-sided [0.656 to 1.692], Standard Error of Mean 0.242

3. Secondary Outcome: Percentage of Participants With Fatigue
Time Frame: Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Month 3 | 89.1
  Month 6 | 38.7
  Month 9 | 19.5
  Month 12 | 13.8

4. Secondary Outcome: Percentage of Participants With Rash
Time Frame: Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Month 3 | 90.6
  Month 6 | 37.9
  Month 9 | 19.5
  Month 12 | 13.8

5. Secondary Outcome: Percentage of Participants With Diarrhea
Time Frame: Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Month 3 | 89.6
  Month 6 | 39.0
  Month 9 | 19.5
  Month 12 | 13.8

6. Secondary Outcome: Percentage of Participants With Rash Based on Severity During the Course of Time
Description: Severity was categorized as Grades 1, 2, 3, 4 and 5. Grade 1= mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2= moderate; minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL). Grade 3= severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4= life-threatening consequences; urgent intervention indicated. Grade 5= death related to adverse event. Only participants that were included in any of the specified categories were reported.
Time Frame: Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Month 3: Grade 1 | 19.2
  Month 3: Grade 2 | 23.1
  Month 3: Grade 3 | 4.4
  Month 6: Grade 1 | 8.1
  Month 6: Grade 2 | 5.7
  Month 6: Grade 3 | 1.0
  Month 9: Grade 1 | 3.6
  Month 9: Grade 2 | 2.3
  Month 12: Grade 1 | 1.8
  Month 12: Grade 2 | 1.6

7. Secondary Outcome: Percentage of Participants With Diarrhea Based on Severity During the Course of Time
Description: as for outcome 6
Time Frame: Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Month 3: Grade 1 | 11.9
  Month 3: Grade 2 | 7.3
  Month 3: Grade 3 | 0.3
  Month 3: Grade 4 | 0.3
  Month 6: Grade 1 | 2.3
  Month 6: Grade 2 | 0.8
  Month 6: Grade 3 | 0.3
  Month 9: Grade 1 | 1.0
  Month 9: Grade 2 | 0.3
  Month 9: Grade 3 | 0.3
  Month 12: Grade 1 | 0.3

8. Secondary Outcome: Percentage of Participants With Fatigue Based on Severity During the Course of Time
Description: as for outcome 6
Time Frame: Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Month 3: Grade 1 | 6.8
  Month 3: Grade 2 | 8.1
  Month 3: Grade 3 | 0.3
  Month 6: Grade 1 | 1.8
  Month 6: Grade 2 | 1.8
  Month 6: Grade 3 | 0.3
  Month 9: Grade 1 | 1.0
  Month 9: Grade 2 | 0.5
  Month 12: Grade 1 | 0.5
  Month 12: Grade 2 | 0.3

9. Secondary Outcome: Percentage of Participants With Dose Modifications by Reason
Description: Dose modification included increase or decreased in the dose of the drug and interrupted dose. Reasons for dose modification included progression, participants' wish, intolerance and others. Only participants that were included in any of the specified categories were reported.
Time Frame: Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Month 3: Increased (other) | 1.0
  Month 6: Increased (other) | 0.8
  Month 9: Increased (other) | 0.3
  Month 12: Increased (participants' wish) | 0.3
  Month 12: Increased (other) | 0.3
  Month 3: Decreased (participants' wish) | 0.3
  Month 3: Decreased (intolerance) | 7.0
  Month 3: Decreased (other) | 0.8
  Month 6: Decreased (participants' wish) | 0.8
  Month 6: Decreased (intolerance) | 1.6
  Month 6: Decreased (other) | 0.3
  Month 9: Decreased (intolerance) | 0.8
  Month 9: Decreased (other) | 0.3
  Month 12: Decreased (intolerance) | 0.5
  Month 3: Interruption (progression) | 0.3
  Month 3: Interruption (intolerance) | 1.8
  Month 3: Interruption (other) | 2.9
  Month 6: Interruption (progression) | 1.0
  Month 6: Interruption (other) | 1.6
  Month 9: Interruption (progression) | 0.5
  Month 9: Interruption (other) | 0.3
  Month 12: Interruption (other) | 0.5

10. Secondary Outcome: Percentage of Participants With Dose Withdrawals by Reason
Description: Reasons for dose withdrawals included progression, participants' wish, intolerance, others and not known. Only participants that were included in any of the specified categories were reported.
Time Frame: Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Month 3: Progression | 34.3
  Month 3: Participants' wish | 2.9
  Month 3: Intolerance | 3.4
  Month 3: Other | 8.3
  Month 3: Not known | 1.0
  Month 6: Progression | 12.7
  Month 6: Participants' wish | 0.5
  Month 6: Intolerance | 0.3
  Month 6: Other | 2.9
  Month 6: Not known | 0.3
  Month 9: Progression | 4.7
  Month 9: Participants' wish | 0.3
  Month 9: Intolerance | 0.3
  Month 9: Other | 1.0
  Month 12: Progression | 2.9

11. Secondary Outcome: Percentage of Participants With Cough by Severity
Description: Severity of cough was categorized as mild, moderate, severe and unknown. Only participants that were included in any of the specified categories in the course of time were reported. Participants with no cough were not included.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Baseline: Mild | 13.8
  Baseline: Moderate | 24.9
  Baseline: Severe | 2.9
  Baseline: Unknown | 1.6
  Month 3: Mild | 15.1
  Month 3: Moderate | 14.5
  Month 3: Severe | 0.3
  Month 3: Unknown | 0.5
  Month 6: Mild | 4.4
  Month 6: Moderate | 3.6
  Month 6: Severe | 0.3
  Month 6: Unknown | 0.5
  Month 9: Mild | 4.7
  Month 9: Moderate | 0.5
  Month 9: Unknown | 0.3
  Month 12: Mild | 1.8
  Month 12: Moderate | 1.3
  Month 12: Severe | 0.3
  Month 12: Unknown | 0.3

12. Secondary Outcome: Percentage of Participants With Dyspnea by Severity
Description: Severity of dyspnea was categorized as mild, moderate, severe, life-threatening and unknown. Only participants that were included in any of the specified categories in the course of time were reported. Participants with no dyspnea were not included.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Baseline: Mild | 16.1
  Baseline: Moderate | 20.3
  Baseline: Severe | 8.1
  Baseline: Unknown | 1.3
  Month 3: Mild | 10.1
  Month 3: Moderate | 17.4
  Month 3: Severe | 4.4
  Month 3: Life-threatening | 0.3
  Month 3: Unknown | 0.8
  Month 6: Mild | 4.7
  Month 6: Moderate | 3.4
  Month 6: Severe | 2.1
  Month 6: Unknown | 0.3
  Month 9: Mild | 3.4
  Month 9: Moderate | 1.0
  Month 9: Severe | 0.5
  Month 9: Unknown | 0.3
  Month 12: Mild | 1.6
  Month 12: Moderate | 0.8
  Month 12: Severe | 0.5
  Month 12: Unknown | 0.3

13. Secondary Outcome: Percentage of Participants With Complete Response (CR), Partial Response (PR) and Stable Disease (SD)
Description: Response rate was observed during the treatment period according to Response Evaluation Criteria in Solid Tumors (RECIST). It consisted of CR, PR, SD and progressive disease (PD). Participants with CR, PR and SD were reported. CR: disappearance of all target lesions (TLs) and non-TLs, with any pathological lymph nodes (whether target or non-target) having a reduction in short axis to less than 10 millimeters (mm). PR: at least a 30 percent (%) decrease in the sum of diameters of TLs, taking as reference the baseline (BL) sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least 20% increase in the sum of diameters of TLs, taking as a reference the smallest sum on study (this included the BL sum if that was the smallest on study). In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm.
Time Frame: Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Month 3: CR | 0.8
  Month 3: PR | 4.9
  Month 3: SD | 25.2
  Month 6: CR | 0.5
  Month 6: PR | 3.1
  Month 6: SD | 14.3
  Month 9: CR | 0.3
  Month 9: PR | 1.6
  Month 9: PD | 10.6
  Month 12: CR | 0.5
  Month 12: PR | 1.6
  Month 12: SD | 8.1

14. Secondary Outcome: Time to Start of Erlotinib Therapy After End of First Line Therapy
Time Frame: Baseline
Population: SAF with number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 373
months | 2.30 [0.03 to 100.39]

15. Secondary Outcome: Percentage of Participants With Remission of CR and PR
Description: Remission was defined as participants with CR or PR. CR: disappearance of all TLs and non-TLs, with any pathological lymph nodes (whether target or non-target) having a reduction in short axis to less than 10 mm. PR: at least a 30% decrease in the sum of diameters of TLs, taking as reference the BL sum diameters.
Time Frame: Months 3, 6, 9, 12
Population: SAF
Measure: Number; unit: percentage of participants
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
percentage of participants
  Month 3 | 5.7
  Month 6 | 3.6
  Month 9 | 1.8
  Month 12 | 2.1

16. Secondary Outcome: Median Progression Free Survival: Overall
Description: Progression-free survival time was defined as the time from the date of first medication to the date of disease progression or death from any cause. If neither progression no death was observed during the study, PFS time was censored at the last day of observation. PD was at least a 20% increase in the sum of diameters of TLs, taking as a reference the smallest sum on study (this included the BL sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm.
Time Frame: From Baseline then every 3 months from Month 3 until disease progression (Maximum follow-up to Month 40)
Population: SAF
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
months | 3.5 [3.2 to 3.9]

17. Secondary Outcome: Median Progression Free Survival: Age
Description: Progression-free survival time was defined as the time from the date of first medication to the date of disease progression or death from any cause. If neither progression nor death was observed during the study, PFS time was censored at the last day of observation. PD was at least a 20% increase in the sum of diameters of TLs, taking as a reference the smallest sum on study (this included the BL sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Median progression-free survival based on the factor of age (65-69, 70-74, 75-79, ≥80 years) were reported.
Time Frame: From Baseline then every 3 months from Month 3 until disease progression (Maximum follow-up to Month 40)
Population: SAF
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
months
  65-69 years | 3.257 [2.632 to 3.914]
  70-74 years | 3.388 [2.763 to 4.079]
  75-79 years | 5.033 [3.717 to 6.382]
  ≥ 80 years | 2.928 [2.039 to 3.750]
Statistical Analysis 1: Comparison: NSCLC Elderly Participants; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.895, Wald Chi-Squares; Hazard Ratio (HR) = 0.981, 95% CI 2-sided [0.741 to 1.299], Standard Error of Mean 0.143
Statistical Analysis 2: Comparison: NSCLC Elderly Participants; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.022, Wald Chi-Squares; Hazard Ratio (HR) = 0.689, 95% CI 2-sided [0.501 to 0.947], Standard Error of Mean 0.162
Statistical Analysis 3: Comparison: NSCLC Elderly Participants; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.479, Wald Chi-Squares; Hazard Ratio (HR) = 1.162, 95% CI 2-sided [0.767 to 1.759], Standard Error of Mean 0.212

18. Secondary Outcome: Median Progression Free Survival: Gender
Description: Progression-free survival time was defined as the time from the date of first medication to the date of disease progression or death from any cause. If neither progression nor death was observed during the study, PFS time was censored at the last day of observation. PD was at least a 20% increase in the sum of diameters of TLs, taking as a reference the smallest sum on study (this included the BL sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Median progression-free survival based on the factor of gender (male and female) were reported.
Time Frame: From Baseline then every 3 months from Month 3 until disease progression (Maximum follow-up to Month 40)
Population: SAF
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
months
  Male | 3.355 [2.993 to 3.750]
  Female | 4.046 [3.257 to 5.888]
Statistical Analysis 1: Comparison: NSCLC Elderly Participants; Comparison between female and male was reported. Parameter estimates, standard errors, Wald Chi-Squares, p-values, hazard ratios and confidence limits were based on a univariate Cox regression with factor gender; Test type: Superiority or Other; p = 0.015, Wald Chi-Squares; Hazard Ratio (HR) = 0.732, 95% CI 2-sided [0.569 to 0.941], Standard Error of Mean 0.129

19. Secondary Outcome: Median Progression Free Survival: Smoking Status
Description: Progression-free survival time was defined as the time from the date of first medication to the date of disease progression or death from any cause. If neither progression nor death was observed during the study, PFS time was censored at the last day of observation. PD was at least a 20% increase in the sum of diameters of TLs, taking as a reference the smallest sum on study (this included the BL sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Median progression-free survival based on the factor of smoking status (smoker, non-smoker and ex-smoker) were reported.
Time Frame: From Baseline then every 3 months from Month 3 until disease progression (Maximum follow-up to Month 40)
Population: SAF
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
months
  Smoker | 3.454 [2.928 to 4.572]
  Non-smoker | 5.526 [3.849 to 10.855]
  Ex-smoker | 2.993 [2.566 to 3.487]
Statistical Analysis 1: Comparison: NSCLC Elderly Participants; Comparison between ex-smoker and non-smoker was reported. Parameter estimates, standard errors, Wald Chi-Squares, p-values, hazard ratios and confidence limits were based on a univariate Cox regression with factor smoking; Test type: Superiority or Other; p = 0.000, Wald Chi-Squares; Hazard Ratio (HR) = 1.902, 95% CI 2-sided [1.402 to 2.582], Standard Error of Mean 0.156
Statistical Analysis 2: Comparison: NSCLC Elderly Participants; Comparison between smoker and non-smoker was reported. Parameter estimates, standard errors, Wald Chi-Squares, p-values, hazard ratios and confidence limits were based on a univariate Cox regression with factor smoking; Test type: Superiority or Other; p = 0.002, Wald Chi-Squares; Hazard Ratio (HR) = 1.786, 95% CI 2-sided [1.248 to 2.557], Standard Error of Mean 0.183

20. Secondary Outcome: Median Progression Free Survival: Best Response to Prior Chemotherapy
Description: Progression-free survival time was defined as the time from the date of first medication to the date of disease progression or death from any cause. If neither progression nor death was observed during the study, PFS time was censored at the last day of observation. PD was at least a 20% increase in the sum of diameters of TLs, taking as a reference the smallest sum on study (this included the BL sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm.
Time Frame: From Baseline then every 3 months from Month 3 until disease progression (Maximum follow-up to Month 40)
Population: Data for best response to prior chemotherapy could not be collected, as it was not recorded in the Case Report Form (CRF), hence, the analysis could not be performed.
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 0

21. Secondary Outcome: Median Overall Survival: Overall
Description: Overall Survival was defined as the time from the date of first medication to the date of death from any cause. If death was not observed during the study, survival time was censored at the last day of observation (latest at the end of study after one year). Overall Survival was analyzed by means of Kaplan-Meier Methods.
Time Frame: From Baseline then every 3 months from Month 3 until death (Maximum follow-up to Month 40)
Population: SAF
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
months | 7.1 [6.0 to 7.9]

22. Secondary Outcome: Median Overall Survival: Gender
Description: Overall Survival was defined as the time from the date of first medication to the date of death from any cause. If death was not observed during the study, survival time was censored at the last day of observation (latest at the end of study after one year). Overall Survival was analyzed by means of Kaplan-Meier Methods. Median survival based on the factor of gender (male and female) were reported.
Time Frame: From Baseline then every 3 months from Month 3 until death (Maximum follow-up to Month 40)
Population: SAF
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
months
  Male | 6.283 [5.526 to 7.467]
  Female | 8.125 [6.349 to 12.237]
Statistical Analysis 1: Comparison: NSCLC Elderly Participants; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.027, Wald Chi-Squares; Hazard Ratio (HR) = 0.717, 95% CI 2-sided [0.535 to 0.962], Standard Error of Mean 0.150

23. Secondary Outcome: Median Overall Survival: Smoking Status
Description: Overall Survival was defined as the time from the date of first medication to the date of death from any cause. If death was not observed during the study, survival time was censored at the last day of observation (latest at the end of study after one year). Overall Survival was analyzed by means of Kaplan-Meier Methods. Median survival based on the factor of smoking status (smoker, non-smoker and ex-smoker) were reported.
Time Frame: From Baseline then every 3 months from Month 3 until death (Maximum follow-up to Month 40)
Population: SAF
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 385
months
  Smoker | 6.612 [5.329 to 8.388]
  Non-smoker | 11.184 [7.928 to NA] — Upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
  Ex-smoker | 5.855 [5.033 to 7.270]
Statistical Analysis 1: Comparison: NSCLC Elderly Participants; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.000, Wald Chi-Squares; Hazard Ratio (HR) = 1.935, 95% CI 2-sided [1.362 to 2.749], Standard Error of Mean 0.179
Statistical Analysis 2: Comparison: NSCLC Elderly Participants; [analysis description as in outcome 19, analysis 2]; Test type: Superiority or Other; p = 0.003, Wald Chi-Squares; Hazard Ratio (HR) = 1.882, 95% CI 2-sided [1.239 to 2.859], Standard Error of Mean 0.213

24. Secondary Outcome: Median Overall Survival: Best Response to Prior Chemotherapy
Description: as for outcome 21
Time Frame: From Baseline then every 3 months from Month 3 until death (Maximum follow-up to Month 40)
Population: Data for best response to prior chemotherapy could not be collected, as it was not recorded in the CRF, hence, the analysis could not be performed.
Arm/Group | NSCLC Elderly Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to Month 40 (Maximum follow-up)
Description: SAF.
Arm/Group | NSCLC Elderly Participants
Serious Adverse Events (participants affected / at risk) | 79/385
Other Adverse Events (participants affected / at risk) | 135/385
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NSCLC Elderly Participants (N=385)
Anaemia (Blood and lymphatic system disorders) | 4
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Disease progression (General disorders) | 2
Fatigue (General disorders) | 2
General physical health deterioration (General disorders) | 6
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Furuncle (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Rash pustular (Infections and infestations) | 4
Sepsis (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
C-reactive protein increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Motor dysfunction (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Reproductive system and breast disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 10
Swelling face (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NSCLC Elderly Participants (N=385)
Diarrhoea (Gastrointestinal disorders) | 52
Fatigue (General disorders) | 41
Cough (Respiratory, thoracic and mediastinal disorders) | 30
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36
Rash (Skin and subcutaneous tissue disorders) | 84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.